CLINICAL TRIAL: NCT05206604
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, VEHICLE-CONTROLLED, FIRST-IN-HUMAN, MULTIPLE-DOSE STUDY, TO INVESTIGATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS, OF TOPICALLY ADMINISTERED PF-07295324 AND PF-07259955, IN HEALTHY ADULT PARTICIPANTS
Brief Title: A First-in-human Study of Multiple Doses of Topically Administered PF-07295324 and PF-07259955
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: C4711001
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07295324 (Experimental): Ointment
  Interventions: Drug: PF-07295324
- PF-07259955 (Experimental): Cream
  Interventions: Drug: PF-07259955

INTERVENTIONS:
Drug: PF-07295324 — Ointment
  Arms: PF-07295324
Drug: PF-07259955 — Cream
  Arms: PF-07259955

SUMMARY:
The purpose of the study is to evaluate the safety, (local and systemic) tolerability, and pharmacokinetics following multiple doses of topically applied, maximum feasible formulations of PF-07295324 (0.12% w/w) or PF-07259955 (2% w/w), on approximately 20% body surface area (BSA), in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

Age and Sex:

1. Healthy (except obese) female participants of non-childbearing potential and/or male participants, at the time of screening, must be 18 to 60 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Male and female of non-child bearing potential participants, who are healthy as determined by medical evaluation including medical history, physical examination, vital assessments, 12 lead ECGs, and laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

   Weight:
4. Body mass index (BMI) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICD and the protocol.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, immunological/rheumatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Participants who have any visible skin damage or skin condition (eg sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations) in or around the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction.
3. Participants who have a history of or have active AD/eczema/urticaria.
4. Evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB) as defined by both of the following:

   * A positive QuantiFERON TB Gold In-tube or equivalent test (QFT).
   * History of either untreated or inadequately treated latent or active TB infection, or current treatment for the same.
5. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed. As an exception a positive HBsAb test due to hepatitis B vaccination is permissible.
6. Have a history of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 1.
7. A history (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
8. Acute disease state (unstable medical condition such as nausea, vomiting, fever or diarrhea, etc) within 7 days of Day 1.
9. Have any malignancies or have a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin.
10. Have a first-degree relative with hereditary immunodeficiency.
11. A history of any lymphoproliferative disorder (such as Epstein Barr Virus [EBV] -related lymphoproliferative disorder), history of lymphoma, leukemia, malignancies or signs and symptoms suggestive of current lymphatic disease.
12. Have undergone significant trauma or major surgery within 4 weeks of screening.
13. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg. Contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

    Prior/Concomitant Therapy:
14. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention. (Refer to Section 6.8 Concomitant Therapy for additional details).
15. Participants who are vaccinated with vaccines that have live components (or live attenuated vaccines) within the 6 weeks prior to the first dose of PF-07295324/vehicle or PF-07259955/vehicle or who are expected to be vaccinated during treatment or during follow-up period.

    NOTE regarding COVID vaccines with authorization or approval for emergency use:

    There is no requirement for washout of COVID vaccines prior to the first dose of PF-07295324/vehicle or PF-07259955/vehicle if the vaccine is not live attenuated (eg, mRNA, utilizing a viral vector,inactivated virus).There is no protocol-specified requirement for the interruption of IP dosing prior to or after vaccination if the COVID vaccine is not live attenuated.
16. Participants in any cohort of this study can only be randomized and receive the IP in only 1 cohort of this study.

    Prior/Concurrent Clinical Study Experience:
17. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).

    Diagnostic Assessments:
18. A positive urine drug test.
19. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
20. Baseline 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
21. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.5 × upper limit of normal (ULN);
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

    Other Exclusions:
22. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
23. Use of tobacco/nicotine containing products more than 5 cigarettes/day.
24. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
25. History of serious adverse reactions or hypersensitivity to any topical drug; or known allergy to any of the test product(s) or any components in the test product(s) or history of hypersensitivity; or allergic reactions to any of the study preparations as described in the PF-07295324 IB and PF-07259955 IB.
26. Not willing to refrain from shaving, the use of depilatories or other hair-removal activities, antiperspirants, lotions, skin creams, fragrances or perfumes, or body oils (eg, baby oil; coconut oil), use of hair products, hair gels, and hair oil in the treatment areas for 48 hours prior to admission to the CRU and for the duration of the stay in the CRU.
27. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
28. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4711001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-four participants were enrolled in the study, with 6 participants assigned to each of the 4 cohorts. All 24 participants were treated: 23 completed the study and 1 discontinued from the study due to non-compliance with study intervention.
Groups:
- Cohort 1 PF-07295324 0.12% Ointment Twice Daily (BID): Healthy participants in Cohort 1 randomized to active received 0.12% PF-07295324 ointment BID on approximately 20% body surface area (BSA) or 4000 cm^2 of skin area for 10 days.
- Cohort 1 PF-07295324 Vehicle Ointment BID: Healthy participants in Cohort 1 randomized to vehicle received vehicle ointment BID on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Cohort 2 PF-07259955 2% Cream BID: Healthy participants in Cohort 2 randomized to active received 2% PF-07259955 cream BID on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Cohort 2 PF-07259955 Vehicle Cream BID: Healthy participants in Cohort 2 randomized to vehicle received vehicle cream BID on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Cohort 3 PF-07295324 0.12% Ointment BID: Healthy participants in Cohort 3 randomized to active received 0.12% PF-07295324 ointment BID on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Cohort 3 PF-07295324 Vehicle Ointment BID: Healthy participants in Cohort 3 randomized to vehicle received vehicle ointment BID on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Cohort 4 PF-07295324 0.12% Ointment Once Daily (QD): Healthy participants in Cohort 4 randomized to active received 0.12% PF-07295324 ointment QD on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Cohort 4 PF-07295324 Vehicle Ointment QD: Healthy participants in Cohort 4 randomized to vehicle received vehicle ointment QD on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
Period: Overall Study
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment Twice Daily (BID) | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment Once Daily (QD) | Cohort 4 PF-07295324 Vehicle Ointment QD
Started | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
Received Treatment | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
Completed | 4 | 2 | 4 | 2 | 4 | 1 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of the study intervention.
Groups:
- Cohort 1 PF-07295324 0.12% Ointment BID: Healthy participants in Cohort 1 randomized to active received 0.12% PF-07295324 ointment BID on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Cohort 4 PF-07295324 0.12% Ointment QD: Healthy participants in Cohort 4 randomized to active received 0.12% PF-07295324 ointment QD on approximately 20% BSA or 4000 cm^2 of skin area for 10 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD | Cohort 4 PF-07295324 Vehicle Ointment QD | Total
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2 | 24
Age, Customized [Number; unit: Participants]
  18 - 44 Years | 2 | 2 | 3 | 0 | 3 | 1 | 2 | 2 | 15
  45 - 60 Years | 2 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 4
  Male | 4 | 2 | 4 | 1 | 3 | 1 | 3 | 2 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 11
  Black or African American | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 10
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Multiracial | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation where participant administered a product; the event did not need to have a causal relationship with the treatment. A SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and non-serious AEs. Treatment-related AEs and SAEs were determined by the investigator.
Time Frame: Baseline up to the end of follow up (ie, up to 44 days)
Population: All participants randomly assigned to study intervention and who are applied at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD | Cohort 4 PF-07295324 Vehicle Ointment QD
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
Participants
  Participants with AEs | 3 | 1 | 1 | 1 | 3 | 2 | 2 | 0
  Participants with treatment-related AEs | 3 | 1 | 1 | 0 | 3 | 1 | 1 | 0
  Participants with SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Hematology parameters included hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet and white blood cell count, total neutrophils, eosinophils, monocytes, basophils, reticulocytes, and lymphocytes. Chemistry parameters included blood urea nitrogen, creatinine, glucose (fasting), calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein. Urine parameters included pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy. Only those categories in which at least 1 participant had abnormal data were reported.
Time Frame: At screening, admission (Day -1), on Days 5, 7, 10, at discharge (Day 12), and at early termination if applicable
Population: All participants randomly assigned to study intervention and who are applied at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD | Cohort 4 PF-07295324 Vehicle Ointment QD
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
Participants
  Neutrophils <0.8*lower limit of normal (LLN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophils/Leukocytes <0.8*LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Eosinophils/Leukocytes >1.2*upper limit of normal (ULN) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Monocytes/Leukocytes >1.2*ULN | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0
  Urate >1.2*ULN | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Potassium >1.1*ULN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Bicarbonate < 0.9*LLN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  URINE Bilirubin >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Leukocyte Esterase >=1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for abnormality in vital signs: supine pulse rate <40 beats per minute (bpm) or >120 bpm; supine diastolic blood pressure (DBP) <50 mmHg, maximum increase or decrease from baseline of >=20 mmHg; supine systolic blood pressure (SBP) <90 mmHg, maximum increase or decrease from baseline of >=30 mmHg. Baseline was defined as the last measurement prior to the first dosing. Vital sign abnormalities reported for at least 1 participant are presented here.
Time Frame: At screening, on Days 1, 2, 5, 7, 10, 11, at discharge (Day 12), and at early termination if applicable
Population: All participants randomly assigned to study intervention and who are applied at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD | Cohort 4 PF-07295324 Vehicle Ointment QD
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
Participants
  Systolic blood pressure decrease >=30 mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic blood pressure increase >=20 mmHg | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Diastolic blood pressure decrease >=20 mmHg | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Findings
Description: ECG abnormalities criteria included: 1) maximum QTc interval adjusted according Fridericia formula (QTcF) (msec): 450<= QTcF <480, 480<= QTcF <500, and QTcF >=500; QTcF maximum increase from baseline (msec): 30<= change <60, and change >=60; 2) maximum PR interval (msec): >=300; PR increase from baseline (msec): baseline >200 with 25% increase at maximum, baseline <=200 with 50% increase at maximum; 3) maximum QRS (msec): >=140; QRS increase from baseline (msec) >=50%. Baseline was defined as the average of the last triplicate measurement prior to the first dosing. ECG abnormalities reported for at least 1 participant are presented here.
Time Frame: At screening, on Days 1, 2, 5, 7, 10, 11, at discharge (Day 12), and at early termination if applicable
Population: All participants randomly assigned to study intervention and who are applied at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD | Cohort 4 PF-07295324 Vehicle Ointment QD
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Skin Irritation Assessments Using Draize Scoring
Description: Application site toleration was assessed by Draize scoring. Draize scores were defined as: 0 = No reaction visible, 1 = Trace reaction - barely perceptible pinkness, 2 = Mild reaction - readily visible pinkness, 3 = Moderate reaction - definite redness, 4 = Strong to severe reaction - very intense redness. Participants with at least 1 instance of Draize score >0 were listed.
Time Frame: Screening up to Day 12 or early termination if applicable
Population: All participants randomly assigned to study intervention and who are applied at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD | Cohort 4 PF-07295324 Vehicle Ointment QD
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 2 | 4 | 2
Participants
  Draize Score = 0 | 2 | 2 | 4 | 2 | 4 | 2 | 4 | 2
  Draize Score = 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Draize Score = 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Draize Score = 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Draize Score = 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07295324 on Days 1 and 10
Description: Cmax was defined as maximum plasma concentration. It was observed directly from data.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: All participants randomly assigned to study intervention who received an application of PF-07295324 and who had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 4 | 4 | 4
ng/mL
  Day 1 | 0.0001000 (0) | 0.0001000 (0) | 0.0001000 (0)
  Day 10 | 0.001655 (19579) | 0.001502 (13373) | 0.002006 (40943)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07295324 on Days 1 and 10
Description: Tmax was defined as time to reach maximum observed plasma concentration. It was observed directly from data.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: All participants randomly assigned to study intervention who received an application of PF-07295324 and who had at least 1 of the PK parameters of interest calculated. In "overall number of participants analyzed", the total number of participants in each treatment group was presented, and in "number analyzed", the number of participants contributing to the data was presented.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 2 | 2 | 2
hour
  Day 1: number analyzed (Participants) | 0 | 0 | 0
  Day 10 | NA [4.00 to 6.00] — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful median when sample size was less than 3. | NA [0.000 to 8.02] — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful median when sample size was less than 3. | NA [4.00 to 8.00] — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful median when sample size was less than 3.

8. Secondary Outcome: Area Under the Concentration-Time Profile From Time Zero to the Dosing Interval Tau (AUCtau) of PF-07295324 on Days 1 and 10
Description: AUCtau was defined as area under the plasma concentration-time profile from time zero to time tau, the dosing interval. tau = 12 hours for BID dosing cohorts and tau = 24 hours for QD dosing cohorts.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 4 | 4 | 4
ng*hr/mL
  Day 1 | 0.0001000 (0) | 0.0001000 (0) | 0.0001000 (0)
  Day 10: number analyzed (Participants) | 3 | 2 | 3
  Day 10 | 0.001262 (1539186) | NA (NA) — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful geometric mean and geometric coefficient of variation when sample size was less than 3. | 0.002037 (82741202)

9. Secondary Outcome: Average Plasma Concentration (Cavg) of PF-07295324 on Days 1 and 10
Description: Cavg was defined as average plasma concentration. It was determined by AUCtau/tau; where tau was the dosing interval and AUCtau was area under the plasma concentration-time profile from time zero to time tau, the dosing interval. tau = 12 hours for BID dosing cohorts and tau = 24 hours for QD dosing cohorts.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 3 | 2 | 3
ng/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 0
  Day 10 | 0.0005518 (7950) | NA (NA) — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful geometric mean and geometric coefficient of variation when sample size was less than 3. | 0.0007061 (30808)

10. Secondary Outcome: Pre-Dose Concentration (Ctrough) of PF-07295324 on Days 1 and 10
Description: Ctrough was defined as pre-dose concentration. It was observed directly from data.
Time Frame: Pre-dose on Days 1 and 10
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 4 | 4 | 4
ng/mL
  Day 1 | 0.0001000 (0) | 0.0001000 (0) | 0.0001000 (0)
  Day 10 (0 hour) | 0.00010008 (0) | 0.0003784 (3451) | 0.0004395 (8008)
  Day 10 (12 hour): number analyzed (Participants) | 4 | 4 | 0
  Day 10 (12 hour) | 0.0001000 (0) | 0.0001000 (0) |

11. Secondary Outcome: Observed Accumulation Ratio for Cmax (Rac[Cmax]) of PF-07295324 on Day 10
Description: Rac(Cmax) was defined as observed accumulation ratio for Cmax and was determined by Cmax on Day 10/Cmax on Day 1. Cmax was defined as maximum plasma concentration. Accumulation ratios was not calculated due to Day 1 Cmax values below the limit of quantification.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 6
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Observed Accumulation Ratio for AUCtau (Rac[AUCtau]) of PF-07295324 on Day 10
Description: Rac(AUCtau) was defined as observed accumulation ratio for AUCtau. AUCtau was defined as area under the plasma concentration-time profile from time zero to time tau, the dosing interval. tau = 12 hours for BID dosing cohorts and tau = 24 hours for QD dosing cohorts. Rac[AUCtau] was calculated by AUCtau on Day 10/AUCtau on Day 1 and accumulation ratios was not calculated due to Day 1 AUCtau values below the limit of quantification.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 6
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Terminal Half-Life (t1/2) of PF-07295324 on Day 10
Description: t1/2 was defined as terminal half-life. It was determined by Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve.
Time Frame: On Days 1, 2, 5, 7, 10, 11, 12, and early termination (if applicable) at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: All participants randomly assigned to study intervention who received an application of PF-07295324 and who had at least 1 of the PK parameters of interest calculated. None of the participants had reportable parameter values.
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Apparent Clearance (CL/F) of PF-07295324 on Day 10
Description: CL/F was defined as aparent clearance. It was determined by Dose/AUCtau. AUCtau was area under the plasma concentration-time profile from time zero to time tau, the dosing interval (12 hours for BID cohorts and 24 hours for QD cohorts).
Time Frame: as for outcome 13
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 1 | 0 | 1
L/hr | NA (NA) — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful geometric mean and geometric coefficient of variation when sample size was less than 3. |  | NA (NA) — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful geometric mean and geometric coefficient of variation when sample size was less than 3.

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-07295324 on Day 10
Description: Vz/F was defined as apparant volume of distribution. It was determined by Dose/(AUCtau * kel). AUCtau was area under the plasma concentration-time profile from time zero to time tau, the dosing interval (12 hours for BID cohorts and 24 hours for QD cohorts). kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve.
Time Frame: as for outcome 13
Population: as for outcome 13
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Cmax of PF-07259955 on Days 1 and 10
Description: Cmax was defined as maximum plasma concentration. It was observed directly from data.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: All participants randomly assigned to study intervention who received an application of PF-07259955 and who had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 4
ng/mL
  Day 1 | 0.001161 (16729163)
  Day 10 | 4.942 (42)

17. Secondary Outcome: Tmax of PF-07259955 on Days 1 and 10
Description: Tmax was defined as time to reach maximum observed plasma concentration. It was observed directly from data.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 16
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 4
hour
  Day 1: number analyzed (Participants) | 0
  Day 10 | 8.00 [0.000 to 23.5]

18. Secondary Outcome: AUCtau of PF-07259955 on Days 1 and 10
Description: AUCtau was defined as area under the plasma concentration-time profile from time zero to time tau, the dosing interval. tau = 12 hours for BID dosing cohorts.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 4
ng*hr/mL
  Day 1: number analyzed (Participants) | 3
  Day 1 | 0.0001000 (0)
  Day 10 | 46.48 (38)

19. Secondary Outcome: Cavg of PF-07259955 on Days 1 and 10
Description: Cavg was defined as average plasma concentration. It was determined by AUCtau/tau; where tau was the dosing interval and AUCtau was area under the plasma concentration-time profile from time zero to time tau, the dosing interval. tau = 12 hours for BID dosing cohorts.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 4
ng/mL
  Day 1: number analyzed (Participants) | 0
  Day 10 | 3.873 (38)

20. Secondary Outcome: Ctrough of PF-07259955 on Days 1 and 10
Description: Ctrough was defined as pre-dose concentration. It was observed directly from data.
Time Frame: Pre-dose on Days 1 and 10
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 4
ng/mL
  Day 1 | 0.0001000 (0)
  Day 10 | 4.077 (41)

21. Secondary Outcome: Rac(Cmax) of PF-07259955 on Day 10
Description: Rac(Cmax) was defined as observed accumulation ratio for Cmax and was determined by Cmax on Day 10/Cmax on Day 1. Cmax was defined as maximum plasma concentration.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 1
ratio | NA (NA) — Per the statistical analysis plan, summary statistics were not presented if fewer than 3 participants had reportable parameter values. Data were considered not sufficient to calculate scientifically meaningful geometric mean and geometric coefficient of variation when sample size was less than 3.

22. Secondary Outcome: Rac(AUCtau) of PF-07259955 on Day 10
Description: Rac(AUCtau) was defined as observed accumulation ratio for AUCtau. AUCtau was defined as area under the plasma concentration-time profile from time zero to time tau, the dosing interval. tau = 12 hours for BID dosing cohorts. Accumulation ratios was not calculated due to Day 1 AUCtau values below the limit of quantification.
Time Frame: On Days 1 and 10 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after application
Population: as for outcome 16
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 0

23. Secondary Outcome: t½ of PF-07259955 on Day 10
Description: as for outcome 13
Time Frame: as for outcome 13
Population: All participants randomly assigned to study intervention who received an application of PF-07259955 and who had at least 1 of the PK parameters of interest calculated. None of the participants had reportable parameter values.
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 0

24. Secondary Outcome: CL/F of PF-07259955 on Day 10
Description: as for outcome 14
Time Frame: as for outcome 13
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 4
L/hr | 3441 (38)

25. Secondary Outcome: Vz/F of PF-07259955 on Day 10
Description: as for outcome 15
Time Frame: as for outcome 13
Population: as for outcome 23
Arm/Group | Cohort 2 PF-07259955 2% Cream BID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to the end of follow up (ie, up to 44 days)
Arm/Group | Cohort 1 PF-07295324 0.12% Ointment BID | Cohort 1 PF-07295324 Vehicle Ointment BID | Cohort 2 PF-07259955 2% Cream BID | Cohort 2 PF-07259955 Vehicle Cream BID | Cohort 3 PF-07295324 0.12% Ointment BID | Cohort 3 PF-07295324 Vehicle Ointment BID | Cohort 4 PF-07295324 0.12% Ointment QD | Cohort 4 PF-07295324 Vehicle Ointment QD
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 3/4 | 1/2 | 1/4 | 1/2 | 3/4 | 2/2 | 2/4 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 PF-07295324 0.12% Ointment BID (N=4) | Cohort 1 PF-07295324 Vehicle Ointment BID (N=2) | Cohort 2 PF-07259955 2% Cream BID (N=4) | Cohort 2 PF-07259955 Vehicle Cream BID (N=2) | Cohort 3 PF-07295324 0.12% Ointment BID (N=4) | Cohort 3 PF-07295324 Vehicle Ointment BID (N=2) | Cohort 4 PF-07295324 0.12% Ointment QD (N=4) | Cohort 4 PF-07295324 Vehicle Ointment QD (N=2)
Application site dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site erythema (General disorders) | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Application site irritation (General disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Application site papules (General disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Application site pruritus (General disorders) | 3 | 1 | 0 | 0 | 3 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT05206604/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT05206604/SAP_001.pdf